CLINICAL TRIAL: NCT02461485
Title: Evaluation of Effects of Fermented Dairy Products Containing Probiotics Alone or in Association With Fibers on Bowel Functions, Constipation Symptoms and Health Related Quality of Life in Adult Subjects With Moderate Constipation: an Exploratory Randomized Double-blind, Controlled Adaptive Study
Brief Title: Effect of a Fermented Milk Product With Probiotics Alone or in Combination With Fibers on Constipation Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NU373
Record Dates: First submitted 2015-04-24; First posted 2015-06-03 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Healthy; Constipation
Keywords: adults; moderate constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1=BOW_01 (Experimental): 1= Fermented Milk Product containing Probiotics
  Interventions: Other: Fermented milk product containing Probiotics
- 2=BOW_01 + fiber C (Experimental): 2= Fermented Milk Product containing Probiotics + Fibers C
  Interventions: Other: Fermented Milk Product containing Probiotics + Fibers C
- 3 =BOW_01 + fiber W (Experimental): 3= Fermented Milk Product containing Probiotics + Fibers W
  Interventions: Other: Fermented Milk Product containing Probiotics + Fibers W
- 4 = Control (Placebo Comparator): 4= Non fermented Milk Product with same color, texture and organoleptic properties as investigational products 1 to 3.
  Interventions: Other: Non fermented Milk Product

INTERVENTIONS:
Other: Fermented milk product containing Probiotics — 2 pots/day during 28 days
  Arms: 1=BOW_01
Other: Fermented Milk Product containing Probiotics + Fibers C — 2 pots/day during 28 days
  Arms: 2=BOW_01 + fiber C
Other: Fermented Milk Product containing Probiotics + Fibers W — 2 pots/day during 28 days
  Arms: 3 =BOW_01 + fiber W
Other: Non fermented Milk Product — 2 pots/day during 28 days
  Arms: 4 = Control

SUMMARY:
First experimental study (Proof Of Concept) to investigate bowel function parameters on which a fermented milk product with probiotics alone or in association with fibers has a potential effect.

ELIGIBILITY:
Main eligibility criteria (non-exhaustive list) are defined as:

* Healthy Caucasian subject of both gender, aged from 18 to 69 years
* Subject with body mass index (BMI) between 18 kg/m2 (bound included) and 30 kg/m2 (bound excluded)
* Subjects with moderate constipation defined according to ROME III adapted criteria.
* Subjects without ongoing or diagnosed gastrointestinal disease or complications.
* Subjects without previous (within one month), ongoing or planned therapy during the study with drugs altering bowel function.
* Subjects without known gluten intolerance, lactose intolerance or allergy to milk proteins.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-10-12 (Actual)

PRIMARY OUTCOMES:
Change in frequency of spontaneous bowel movements by questionnaire at baseline and after 4 weeks. | Baseline and after 4 weeks.
Change in stool consistency (Bristol Stool Scale) at baseline and after 4 weeks. | Baseline and after 4 weeks.
Change in Whole Gut Transit Time (radio-opaque markers) at baseline and during the 4th week. | Baseline and during the 4th week.
Change in fecal bulk (stool weight) at baseline and after 4 weeks. | Baseline and after 4 weeks.
Change in constipation symptoms assessed by questionnaire at baseline and after 2 and 4 weeks. | Baseline and after 2 and 4 weeks. Validated questionnaire.
Evolution of Health related Quality of Life assessed by questionnaire at baseline and after 2 and 4 weeks. | Baseline and after 2 and 4 weeks. Validated questionnaire.
Study product satisfaction by questionnaire after 2 and 4 weeks. | after 2 and 4 weeks.
Adverse events in the week before baseline, at baseline, week 3, 4 and 5. | Evaluation of safety will be assessed with AE and SAE reporting throughout the whole study i.e. day -7 (screening period), day 0 (randomisation), day 15, day 22 and day 29 (end of study)

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland